CLINICAL TRIAL: NCT07034599
Title: Effects of Negative Pressure Ventilation Onto Hemodynamics and Right Ventricular Funktion in Patients After Implantation of a Left Ventricular Assist Device.
Acronym: NPV LVAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karlsburg Hospital (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Matthias Heringlake, Head of department for anesthesiology and critical care, Karlsburg Hospital
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KAIKB 2025-2
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Critical Illness; Heart Failure; LVAD
MeSH Terms: conditions — Critical Illness; Heart Failure | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants negative pressure ventilation and positive pressure ventilation (Experimental)
  Interventions: Device: Negative pressure ventilation; Device: positive pressure ventilation

INTERVENTIONS:
Device: Negative pressure ventilation — All participants are ventilated with negative pressure ventilation first
Device: positive pressure ventilation — All participants are ventilated using positive pressure ventilation after negative pressure ventilation

SUMMARY:
All patients undergoing an implantation of a durable left ventricular assist device and monitored by pulmonary artery catheter showing no adverse events after surgery are included in the study and ventilated for 15 minutes using extra thoracic negative pressure ventilation and usual intrathoracic positive pressure ventilation. Hemodynamics changes between both ventilation modes, especially focussing on right ventricular function and measured by a pulmonary artery catheter, are compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients after implantation of a durable left ventricular assist device

Exclusion Criteria:

* Complication during surgery like bleeding, emergency, inability to fit the cuirass, unavailability of an investigator, unstable condition regarding circulation or ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
RVSWI | one minute
  right ventricular stroke work index

IPD SHARING:
Plan to Share IPD: Undecided